## Comparison of Honey and Povidone-iodine in Wound Healing on Acute Laceration Wounds: A Randomized Controlled Trial Study

NCT03641053

Document Date: September 4, 2017

## PART II: Approval Page to become a Respondent

## APPROVAL PAGE TO BECOME A RESPONDENT (INFORMED CONSENT)

| I, the unde | ersigned | be. | low: |
|-------------|----------|-----|------|
| NT | _ | | |

Name : Age : Address :

(fill in if respondent is under the age of 21 years old) Relation with respondent is parent/guardian of the child:

Name : Age :

Have read the information stated above, or have been read to me. I have had the chance to ask of the information above and every single question of mine has been answered completely. I have understood the procedure of the research that will be executed, alongside the benefits, goals, and also the chance of negative impacts that may arise. I volunteer to participate in this research with no obligations nor force from any parties. I believe that the safety and secrecy of this research's data will be guaranteed, and with this I hereby agree to every data produced in this research to be publicized in any form of oral and written. If in the future there is any difference, then it will be solved by a mutual agreement.

NAME SIGNATURE DATE/MONTH/YEAR

Respondent

Witness 1

Witness 2

## **Head of Research Team:**

Name : Kevin Leonard Survadinata

Address : Timor Raya Road. no. 134, Pasir Panjang,

Kupang, East Nusa Tenggara

Telephone: +62 813 3685 5247

APPROVED BY THE HEALTH
RESEARCH ETHICS COMMITTEE OF
MEDICAL FACULTY OF NUSA
CENDANA UNIVERSITY
September 4, 2017



This document was created with the Win2PDF "print to PDF" printer available at <a href="http://www.win2pdf.com">http://www.win2pdf.com</a>

This version of Win2PDF 10 is for evaluation and non-commercial use only.

This page will not be added after purchasing Win2PDF.

http://www.win2pdf.com/purchase/